CLINICAL TRIAL: NCT05495984
Title: Neuroplasticity in Maternal Opioid Use Disorder (OUD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2000033065
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Evoked Potentials

STUDY DESIGN:
Intervention Model Description: All participants (n=15) will complete Study Visit 1 for the Primary Objective, and Study Visits 2-14 for the Secondary Objective.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Objective: Event-Related Potentials (ERPs) (Experimental): Use ERPs elicited by unknown infant face and cry stimuli to determine whether neural markers translate to maternal mentalization in mothers with opioid use disorder (OUD) at 4-12 months postpartum
  Interventions: Behavioral: ERPs with electroencephalography (EEG)
- Secondary Objective: ERPs + Mothering from the Inside Out (MIO) (Experimental): Use Event-Related Potentials (ERPs) elicited by unknown infant face and cry stimuli to determine whether neural response changes with participation in an evidence-based parenting intervention designed specifically for mothers with OUD: Mothering from the Inside Out (MIO).
  Interventions: Behavioral: ERPs with electroencephalography (EEG); Behavioral: MIO

INTERVENTIONS:
Behavioral: ERPs with electroencephalography (EEG) — E-Prime 2.0 software will present visual and auditory stimuli in an experimental paradigm lasting approximately 30 minutes (ERPs). Visual stimuli will include photographs of color photographs of unfamiliar infants (aged 5- 10 months) balanced for ethnicity (Black/White) and gender (male/female) displaying happy neutral, and sad affective expressions. Auditory stimuli will include 2-second audio clips of high-distress and low-distress infant cries. Experimental procedure: Trials will consist of a central fixation cross (jittered 400-600ms), stimulus presentation (500ms faces, 2000ms cries), and blank screen (1000ms). Continuous electroencephalography (EEG) will be recorded using Net Station 4.2.1. A 128 Ag/Silver Chloride (AgCl) electrode net will be soaked in a warm potassium chloride solution, and net electrodes will be spaced evenly and symmetrically on each participant's head to cover the scalp.
Behavioral: MIO — A 12-week, manualized, individual parenting psychotherapy developed specifically for mothers with addictions administered by the Principal Investigator. It is designed to foster a mother's capacity for mentalization or reflective functioning (RF). MIO is offered in conjunction with standard addiction treatment.
  Arms: Secondary Objective: ERPs + Mothering from the Inside Out (MIO)

SUMMARY:
Opioid use disorder (OUD) remains a major public health problem particularly for mothers in the perinatal period, for whom stress, relapse rates, and risk for overdose are elevated. The perinatal period is characterized by significant neural reorganization that determines outcomes for mothers and infants. OUD is also associated with neural reorganization, specifically neural circuitry implicated in stress regulation and reward processes. Interventions should therefore take advantage of this changing perinatal biology to enhance treatment response by targeting the aberrant neural circuitry compromised by maternal OUD. The investigators have developed and refined an evidence-based intervention for mothers with OUD designed to target these neural mechanisms and enhance the reward of caregiving; however, this has yet to be formally tested. Therefore, the investigators will examine maternal neuroplasticity using high-dense array electroencephalography (EEG) in mothers with OUD in response to our intervention. There will be 1 laboratory visit at pre-treatment, followed by 12 sessions of the evidence-based parenting intervention, and 1 laboratory visit at post-treatment. This study will attempt to validate the importance of taking advantage of the neuroplasticity in the perinatal period to optimize outcomes for mothers with OUD.

DETAILED DESCRIPTION:
This is a study conducted at the Child Study Center (CSC) in the Yale School of Medicine. It involves mothers in treatment for OUD who are caring for infants who are 4-12 months old.

15 mothers will complete 1 study visit, which will last 2.5 hours. It will start with informed consent and then will include demographics, EEG/ERP, a multidimensional assessment of mentalization (a brief self-report questionnaire, a 5-minute speaking task, and a one-hour interview) and several clinical measures (depression, anxiety, stressful life events).

Participants will then complete 12 treatment (Mothering from the Inside Out (MIO)) visits, and 1 post-treatment data collection visit.

Visits 2-13 (1 hour each) consist of participation in Mothering from the Inside Out (MIO).

Visit 14 (2.5 hours) includes participation in the ERP paradigm and the multidimensional assessment of mentalization (a brief self-report questionnaire, a 5-minute speaking task, and a one-hour interview) and several clinical measures (depression, anxiety, stressful life events).

ELIGIBILITY:
Inclusion Criteria:

* Biological mother of infants between 4-months and 12-months of age
* 21-45 years of age at time of recruitment
* Enrolled in substance use treatment and on mediation for opioid use disorder (MOUD).

Exclusion Criteria:

* Incapable of giving informed consent
* Child spends less than 50% of time in mother's custody.
* Non-English-speaking
* Unable to complete the study because of pending legal cases or unable to supply two forms of contact for the purpose of follow-up
* Physiological addiction to a substance that requires detoxification, defined as difficulties with physiological withdrawal from substances (e.g. delirium tremens, shaking, nausea).

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in mothers' Event-related potentials (ERPs) elicited by unknown infant face and cry stimuli | Week 1 and Week 14
  E-Prime 2.0 software will present visual and auditory stimuli in an experimental paradigm lasting approximately 30 minutes. Continuous electroencephalography (EEG) will be recorded using Net Station 4.2.1. Net Station 4.5 will be used to pre-process EEG data (first be digitally filtered, then segmented into 1-second epochs (100ms pre- and 900ms post-stimulus onset). Net Station artifact detection will be set to detect artifact. Spline interpolation will be used to replace channels with artifacts in more than 40% of trials. Ocular Artifact Removal (OAR), using a blink slope threshold of 14µV/ms, will be applied to data for all participants. EEG data will next be re-referenced to the average reference of all electrodes and baseline corrected to the 100ms interval pre-stimulus onset. Lastly, the EEG data will be averaged across stimulus conditions for each participant. The N170, N100, and P300 will be visually inspected in the grand-averaged data and verified for each participant.
Change in maternal mentalization measured by coding of reflective functioning (RF) on the one-hour Parent Development Interview (PDI) | Week 1 and Week 14
  The PDI is a semi-structured interview with 19 questions eliciting a parent's verbal narrative about common emotionally-challenging aspects of parenting. The interview is recorded, transcribed, and each of the 19 responses is rated on a 10-point scale where: a score of 1 indicates complete absence of recognition of mental states (events are described solely in terms of behavior) and scores above 5 indicate increasingly elaborate and sophisticated understanding of how mental states function and influence behavior. Reliable coders assign an Overall Score to the protocol that represents the parent's modal level of response. The PDI requires approximately 60 minutes to complete.
Change in mothers' reflective functioning assessed using the self-report Parental Reflective Functioning Questionnaire (PRFQ) | Week 1 and Week 14
  The PRFQ is an 18-item self-report questionnaire to quantify levels of 3 key components of parental RF: Interest & Curiosity surrounding their child's mental states, Certainty in the recognition of their child's mental states, and Pre-Mentalizing or difficulty in considering the child's mental states. Optimal RF is indicated by higher scores on the interest and curiosity subscale, moderate scores on the certainty subscale, and lower scores on the pre-mentalizing subscale. Participants rate their responses on a 7-point likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). The PRFQ requires approximately 10 minutes to complete.
Change in mothers' certainty about mental states assessed using the self-report Certainty about Mental States Questionnaire (CAMSQ) | Week 1 and Week 14
  The CAMSQ is a psychometrically sound 20-item self-report questionnaire. The CAMSQ assesses two maladaptive variants of subjective certainty about mental states that can be linked to hypomentalizing and hypermentalizing. The CAMSQ yields two subscales representing certainty about one's own metal states, and certainty about others' mental states. Items are scored by taking the mean of item responses (never = 1, almost never = 2, sometimes = 3, half of the time = 4, often = 5, almost always = 6, always = 7). The CAMSQ requires approximately 15 minutes to complete.
Change in mothers' mind-mindedness assessed using the Five-Minute Speech Sample (MM) | Week 1 and Week 14
  On the five-minute speech sample, mothers will be asked to describe their child for five minutes; responses will be recorded, transcribed, and coded using the representational MM coding manual. Descriptions that refer to mental states (e.g., cognitions, emotions, desires, interests) are identified as mind-minded. The frequency of mind-minded comments will be calculated, as will the proportion of mind-minded to non- mind-minded comments, to control for verbosity.

SECONDARY OUTCOMES:
Mothers' baseline substance use assessed using the Addiction Severity Index (ASI-Lite) | Week 1
  This interview characterizes mothers' recent (past 30 day) and lifetime substance use. Seven potential problem areas are assessed: Medical, Employment/Support Status, Alcohol, Drug, Legal, Family/Social, and Psychological. For each area, mothers will be asked to rate the impact of their substance use, using the following scale: (0) Not at all; (1) Slightly; (2) Moderately; (3) Considerably; (4) Extremely. The ASI-Lite requires approximately 15 minutes to complete.
Change in mothers' depression assessed using the Edinburgh Postnatal Depression Scale (EPDS) | Week 1 and Week 14
  The EPDS is a 10-item questionnaire that uses a 4-point Likert scale. Participants are asked to rate the extent to which in the past 7 days they have experienced symptoms such as feeling unhappy, panicky, sad, or tearful. Scores range from 0 to 30, and the threshold for the presence of possible depression is 10. The EPDS requires approximately 5 minutes to complete.
Change in mothers' depression assessed using the Patient Health Questionnaire-2 (PHQ-2) | Week 1 and Week 14
  The PHQ-2 is a brief, 2-item screening tool that asks on a 4-point Likert scale how often over the past two weeks participants have been bothered by little interest or pleasure in doing things and feeling down/depressed/hopeless. Scores range from 0 to 8. The PHQ-2 requires approximately 1 minute to complete.
Change in mothers' anxiety assessed using the Generalized Anxiety Disorder-7 (GAD-7) | Week 1 and Week 14
  The GAD-7 is a brief, 7-item screening tool that asks on a 4-point Likert scale how often over the past two weeks participants have been bothered by symptoms of generalized anxiety (e.g., feeling nervous, worry, difficulty relaxing, restlessness, irritability, etc.) Scores range from 0 to 21. The GAD-7 requires approximately 5 minutes to complete.
Change in mothers' stress assessed using the Parenting Stress Index- Short Form (PSI-SF) | Week 1 and Week 14
  The PSI-SF is a 36-item self-report questionnaire for parents of children who are younger than 12 years of age. Parents are asked to rate their agreement with statements on a 5-point likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The PSI-SF yields a Total Stress score, as well as 3 subscales (each consisting of 12 items): Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. Responses from each item are summed for each subscale and all items are included in the Total Stress score, with higher scores representing higher levels of parenting stress. The PSI-SF requires approximately 15 minutes to complete.
Mothers' experience of childhood maltreatment assessed using the Childhood Trauma Questionnaire (CTQ) | Week 1
  The CTQ is a 28-item self-report questionnaire asking parents to indicate the frequency of their traumatic experiences on a 5-point Likert scale ranging from 1 (never true) to 5 (very often true). The CTQ yields 5 subscales: emotional abuse, physical abuse, sexual abuse, emotional neglect, and physical neglect. Each subscale consists of 5 questions and scores can thus range from 5 to 25. The remaining 3 questions are used to assess participants minimization or denial of their experiences, which would suggest an underreporting of traumatic experiences. The CTQ requires approximately 15 minutes to complete.
Mothers' experience of childhood adversity assessed using the Adverse Childhood Experiences Scale (ACES) | Week 1
  The ACES is a 10-item questionnaire that assesses exposure to various adversities before the age of 18. Participants are asked to indicate whether or not they experienced 10 different kinds of adversities in a dichotomous no/yes format. Scores can thus range from 0 to 10, with higher scores representing exposure to a greater number of types of adversity. The ACES requires approximately 5 minutes to complete.
Change in mothers' internalized stigma assessed using the Brief Opioid Stigma Scale (BOSS) | Week 1 and Week 14
  The BOSS is a 7-item self-report questionnaire that assesses internalized stigma experienced by individuals with an opioid use disorder. Participants respond using a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The BOSS yields 3 subscales: Aware (i.e., awareness of stereotypes), Agree (i.e., agreement with stereotypes), and Harm (i.e., negative impact to self-esteem), with higher scores representing higher levels of internalized stigma. The BOSS requires approximately 5 minutes to complete.
Change in mothers' internalized stigma assessed using the Substance Use Stigma Mechanism Scale (SU-SMS) | Week 1 and Week 14
  The SU-SMS is an 18-item self-report questionnaire that assesses enacted stigma (i.e., experiences of discrimination from others), anticipated stigma (expectations of experiencing discrimination), and internalized stigma (the application of negative beliefs about people with substance use disorders to onesself). Participants respond on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Each subscale yields a score that can range from 6 to 30, with higher scores representing higher levels of stigma. The SU-SMS requires approximately 10 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Lowell, Ph.D., Principal Investigator — Yale University; Helena Rutherford, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Child Studies Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No